CLINICAL TRIAL: NCT07119879
Title: Impact of Climate Change Anxiety on Sinusitis Symptoms and Quality of Life Among Adults With Chronic Rhinosinusitis: A Cross-Sectional Study
Acronym: CLIM-RHINO (Cl
Status: Completed | Type: Observational
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, lecturer, Sinai University
Other Study IDs: IRB00014233-17
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Rhinosinusitis (CRS); Climate Change Anxiety; Quality of Life Impairment
Keywords: SNOT-22; psychosomatic health; environmental stress; quality of life; climate change anxiety; Chronic rhinosinusitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Chronic Rhinosinusitis: This cross sectional includes adult participants (≥18 years) with self-reported or physician-diagnosed chronic rhinosinusitis who completed an online questionnaire assessing climate change anxiety, SNOT-22 scores, and quality of life.

SUMMARY:
This cross-sectional observational study investigates the relationship between climate change anxiety and chronic rhinosinusitis (CRS) symptom severity and quality of life (QoL) in adults. As climate change continues to influence public health, individuals with chronic respiratory diseases may experience worsened symptoms due to heightened psychological stress and perceived environmental instability. The study utilizes standardized instruments including the SNOT-22 (Sino-Nasal Outcome Test), a QoL scale, and a climate change anxiety questionnaire to evaluate associations among these variables.

DETAILED DESCRIPTION:
Climate change has emerged as a major global health concern, with growing recognition of its psychological impacts, including anxiety, distress, and perceived environmental instability. These psychosocial effects may exacerbate symptoms in chronic inflammatory conditions such as Chronic Rhinosinusitis (CRS), a disease characterized by persistent nasal congestion, facial pressure, and impaired quality of life.

This study aims to explore the correlation between self-perceived climate change anxiety and CRS symptom severity and QoL in an adult population. A total of 134 participants with CRS, aged ≥18 years, were recruited to complete an online Arabic-language survey. The survey included demographic information, the SNOT-22 scale, a validated quality of life questionnaire, and a climate change stress scale.

The primary objective is to assess the association between climate change stress and symptom severity (SNOT-22 total score). The secondary objective is to determine the relationship between climate change anxiety and QoL. The study uses Pearson's correlation analysis to examine these associations.

This research introduces a novel psychosomatic dimension to CRS management by highlighting how environmental and psychological stressors may influence disease burden. Results may inform multidisciplinary approaches for patient care, incorporating environmental awareness and mental health support.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following:

Adults aged 18 years or older Self-reported or clinically diagnosed with Chronic Rhinosinusitis (CRS) with symptoms lasting ≥12 weeks Able to read and understand Arabic Able to complete the online questionnaire independently Provided informed consent prior to participation Exclusion Criteria

Participants will be excluded if they meet any of the following:

Diagnosis of severe psychiatric or psychological disorders (e.g., schizophrenia, bipolar disorder) History of major chronic illnesses that may confound outcomes (e.g., cardiovascular disease, cancer, chronic neurological disease) Recent nasal or sinus surgery within the past 3 months Incomplete survey responses that prevent data analysis Participants under 18 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study targets adult individuals (aged ≥18 years) residing in Egypt who have self-reported or medically diagnosed Chronic Rhinosinusitis (CRS) with symptom duration of at least 12 weeks. Participants were required to read and understand Arabic in order to complete a structured online questionnaire. Recruitment was conducted electronically through convenience sampling via social media and academic platforms.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Correlation between Climate Change Anxiety and CRS Symptom Severity | Day 1 (Single assessment at time of survey completion)
  Evaluate the relationship between participants' climate change anxiety scores and their chronic rhinosinusitis symptom severity using the SNOT-22 questionnaire.

SECONDARY OUTCOMES:
Correlation between Climate Change Anxiety and Quality of Life | Day 1 (Single assessment at time of survey completion)
  Assess the relationship between climate change anxiety scores and health-related quality of life (QoL) scores among adults with CRS.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai university, Cairo, Egypt